CLINICAL TRIAL: NCT05321056
Title: Exposure Measurements and Interventions for Aerosol Produced by Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, SHENGYU ZHANG, Principal Investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZS-3377
Record Dates: First submitted 2022-03-16; First posted 2022-04-11 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Droplet Transmission
Keywords: Exposure Risk; Digestive Endoscopy; Personal protective equipment
MeSH Terms: interventions — Masks; Ventilators, Mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Mask on model face (Experimental): The mask (surgical mask, respirator) will be worn on the face of the in vitro bionic model.
  Vitamin B2 saline solution of the same dose will be dripped into each patient's mouth before EGD examination, as a fluorescent tracer.
  Interventions: Device: masks (surgical mask, respirator)
- Control group: No mask on model face (No Intervention): No mask (surgical mask, respirator) will be worn on the face of the in vitro bionic model.
  Vitamin B2 saline solution of the same dose will be dripped into each patient's mouth before EGD examination, as a fluorescent tracer.

INTERVENTIONS:
Device: masks (surgical mask, respirator) — The mask (surgical mask, respirator) will be worn on the face of the in vitro bionic model in the procedure room for measuring droplet exposure.
  Arms: Intervention group: Mask on model face

SUMMARY:
Study objective: To clarify the risk of exposure to the exhaled aerosol droplets from patients for medical staffs during digestive endoscopy via labelling the oral mucosa with vitamin B2 solution, and evaluate the protective efficacy of personal protective equipment.

Study design: This is a prospective randomized controlled study.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study. Patients who meet the inclusion criteria and do not meet the exclusion criteria are recruited for this trial. They will be randomly divided into the control group and the intervention group (A total of 70 subjects, and 35 per group based on calculation of sample size). The in vitro bionic model next to the doctor simulated a medical staff, which is printed via the stereolithographic appearance 3D printing technique following the morphological structure data of human face and airway obtained by processing CT images, will either wear a mask or not, depending on the intervention group (in the intervention group, in vitro model wears personal protective equipment). Before starting the esophagogastroduodenoscopy (EGD) under anesthesia, vitamin B2 saline solution (vitamin B2 dosage determined by the suggested daily nutrient uptake in China) is dripped in their mouths. When the examination is finished, the dosage of facial mucosa deposition and airway inhalation of the in vitro model is quantified as a cumulative droplet mass (μg) over all the exposure time. The deposited droplets are collected by wiping method, and the inhaled droplets are sampled by a solution-based sampler (SKC, U.S.A.). The dosage is detected by the Fluoro Max-4® fluorophotometer (HORIBA, Japan). By comparing and analyzing the results of the two intervention groups, the researchers try to evaluate the risk of exposure under the personal protective equipment and assess the effectiveness of it.

ELIGIBILITY:
Inclusion Criteria:

* During the study period, patients who were treated in the digestive endoscopy center of Peking Union Medical College Hospital and planned to undergo digestive endoscopy. Age and gender are not limited temporarily.

Exclusion Criteria:

* Patients who have ever been allergic to the medical non-toxic fluorescent agent ( vitamin B2 saline solution).
* Patients who received anti-tumor therapy during the period of digestive endoscopy.
* Patients with poor general conditions, including severe cardiopulmonary diseases, coagulation disorders, or a total of platelet less than 50*10^9/L.
* Patients with structural pulmonary disease (chronic obstructive pulmonary disease, asthma, etc.) or airway/pulmonary surgery history
* Patients with intolerance or contraindications to digestive endoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Dosage of in vitro model airway inhalation of patient's exhaled droplets | one year
  After EGD examination, the dosage of airway inhalation of the in vitro model is quantified as a cumulative droplet mass (μg) over all the exposure time. The deposited droplets are collected by wiping method, and the inhaled droplets are sampled by a solution-based sampler (SKC, U.S.A.). The dosage is detected by the Fluoro Max-4® fluorophotometer (HORIBA, Japan).

SECONDARY OUTCOMES:
Dosage of in vitro model facial mucosa deposition of patient's exhaled droplets | one year
  After EGD examination, the dosage of facial mucosa deposition of the in vitro model is quantified as a cumulative droplet mass (μg) over all the exposure time. The deposited droplets are collected by wiping method, and the inhaled droplets are sampled by a solution-based sampler (SKC, U.S.A.). The dosage is detected by the Fluoro Max-4® fluorophotometer (HORIBA, Japan).

CONTACTS AND LOCATIONS:
Overall Officials: Shengyu Zhang, M.D., Study Director — Peking Union Medical College Hospital; Zhiyu Yan, M.D. Program, Principal Investigator — Peking Union Medical College Hospital; Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Yan Z, Zhang Y, Wu X, Liu L, Yang A, Duan M. Protocol of a randomised controlled trial to assess medical staff's inhalation exposure to infectious particles exhaled by patients during oesophagogastroduodenoscopy and the efficacy of surgical masks in this context. BMJ Open. 2023 Feb 28;13(2):e068291. doi: 10.1136/bmjopen-2022-068291. PMID 36854596